CLINICAL TRIAL: NCT03263117
Title: SEGA - SEdation Versus General Anesthesia for Endovascular Therapy in Acute Ischemic Stroke - a Randomized Comparative Effectiveness Trial.
Brief Title: SEdation Versus General Anesthesia for Endovascular Therapy in Acute Ischemic Stroke
Acronym: SEGA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Stryker Neurovascular (Industry)
Responsible Party: Principal Investigator, Peng Roc Chen, MD, Professor in Neurosurgery, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-MS-17-0436
Record Dates: First submitted 2017-08-16; First posted 2017-08-28 (Actual); Results first posted 2024-09-05 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-09

CONDITIONS: Stroke
Keywords: Acute stroke; Cerebral Stroke
MeSH Terms: conditions — Stroke | interventions — Anesthesia, General

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sedation (Active Comparator): The protocol does not specify a particular combination of drugs that must be used for sedation. The choice of specific drugs and dosages for achieving sedation will be up to the anesthesiologist.
  Interventions: Drug: Sedation; Procedure: Intra-arterial Thrombectomy
- General Anesthesia (Active Comparator): The protocol does not specify a particular combination of drugs that must be used for general anesthesia. The choice of specific drugs and dosages for achieving general anesthesia will be up to the anesthesiologist.
  Interventions: Drug: General Anesthesia (GA); Procedure: Intra-arterial Thrombectomy

INTERVENTIONS:
Drug: Sedation — The protocol does not specify a particular combination of drugs that must be used for sedation.
  The most common drugs utilized for sedation and wide dosing ranges are included in the protocol (i.e., sedation will be provided under the supervision of an anesthesiologist and may use a combination of fentanyl, midazolam, dexmedetomidine infusion (with or without loading dose), and/or low-dose propofol by intermittent bolus or infusion); however, the choice of specific drugs and dosages for achieving conscious sedation or general anesthesia will not be specified by the protocol but will be up to the anesthesiologist.
  Arms: Sedation
Drug: General Anesthesia (GA) — The protocol doesn't specify drugs that must be used for GA, the choice of drugs and dosages for achieving general anesthesia will not be specified by the protocol but will be up to the anesthesiologist.
  The most common drugs utilized for GA and wide dosing ranges included in the protocol are (GA will be provided under the supervision of an anesthesiologist and induction of anesthesia may be achieved with propofol and/or etomidate; muscle paralysis may be achieved with succinylcholine or non-depolarizing paralytic (rocuronium or vecuronium); and adjuvant lidocaine and fentanyl; if intravenous maintenance of anesthesia is used, it may be achieved by propofol infusion at 50 to 150 mcg/kg/min with redosing of non-depolarizing paralytic and fentanyl as needed; if inhalational maintenance of anesthesia is used it will be achieved with sevoflurane 1% to 2% or desflurane 3% to 6% end-tidal concentration with redosing of non-depolarizing paralytic and fentanyl as needed)
  Arms: General Anesthesia
Procedure: Intra-arterial Thrombectomy — The first line therapeutic embolectomy device should be a stent retriever. Additional Endovascular therapies including, but not limited to, intra- or extracranial angioplasty ± stenting; antithrombotics (oral, IV or IA antiplatelets or anticoagulants) intra-arterial thrombolytics; are left to the decision of the local treatment team.
  Other Names: Endovascular Therapy

SUMMARY:
Objectives:

This study aims to estimate overall treatment benefit (improvement in disability) among acute ischemic stroke patients that are randomized to General Anesthesia (GA) compared with Sedation (CS) during endovascular therapy. Assess safety (as measured by incidence of symptomatic intracranial hemorrhage); rates of Endovascular therapy (EVT) procedural complications, reperfusion; and quality of life.

Hypothesis:

GA during EVT for acute ischemic stroke improves functional outcomes at 90 days compared to sedation.

ELIGIBILITY:
Inclusion Criteria:

1. Acute ischemic stroke due to large intracranial vessel occlusion demonstrated on CT-angiography in the following anterior circulation locations that will be treated by endovascular therapy (EVT):

   1. Internal Carotid Artery (terminal "T" or "L-type"- occlusion)
   2. Middle Cerebral Artery (MCA) M1 or proximal M2
   3. Anterior Cerebral Artery (ACA) A1 or proximal A2

      * Patients who receive IV-tPA thrombolysis are eligible provided the drug was delivered within 4.5 hours of stroke onset or last seen normal and in accordance with local hospital standard of care.
2. Ages 18-90.
3. National Institute of Health Stroke Scale (NIHSS) score 6-30
4. Time of from stroke symptom onset of last seen normal to start of EVT (defined as groin puncture) ≤ 16 hours.
5. Limited infarct core, as defined below and adapted from the 2018 American Heart Association guidelines

   1. For patients presenting ≤ 6 hours from time of symptom onset or last seen normal, Alberta Stroke Program Early Computed Tomography Score (ASPECTS) ≥ 6
   2. For patients presenting > 6 hours and ≤ 16 hours from time of symptom onset or last seen normal, they must satisfy EITHER ONE of the two following criteria:

   i. Ischemic core by CT Perfusion or MRI/MR Perfusion < 70 mL, a ratio of volume of penumbral tissue to infarct core of ≥ 1.8, and and absolute volume of penumbral tissue of ≥ 15 mL OR ii. For patients with NIHSS ≥ 10, infarct core of < 31 mL by CT Perfusion or MRI; For patients with NIHSS ≥ 20, infarct core < 51 mL.
6. Subject willing/able to return for protocol required follow up visits.
7. No significant pre-stroke disability (modified Rankin Score must be ≤ 2).
8. Females of childbearing potential must have a negative serum or urine pregnancy test.
9. Patient or patient's legally authorized representative has given Informed Consent according to Good Clinical Practices (GCP) and/or local IRB policies.

Exclusion Criteria:

1. Coma on admission (Glasgow Coma Scale <8), need for intubation upon ED arrival, or transferred patients who present previously intubated.
2. Severe agitation or seizures on admission that preclude safe vascular access.
3. Loss of airway protective reflexes and/or vomiting on admission.
4. Predicted or known difficult airway.
5. Pre-existing neurological or psychiatric disease that would confound the neurological or functional evaluations, e.g. dementia.
6. Presumed septic embolus, or suspicion of bacterial endocarditis
7. Currently participating or has participated in any investigational drug or device study within 30 days.
8. Inability to follow-up for 90-day assessment.
9. Known history of allergy to anesthesia drugs.
10. Known history or family history of malignant hyperthermia

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2023-04-22 (Actual); Study Completion 2023-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peng Roc Chen, MD, Study Chair — The University of Texas Health Science Center, Houston; Andrew Barreto, MD, Principal Investigator — The University of Texas Health Science Center, Houston; Carlos Artime, MD, Principal Investigator — The University of Texas Health Science Center, Houston; Sunil Sheth, MD, Principal Investigator — The University of Texas Health Science Center, Houston; Sean Savitz, MD, Principal Investigator — The University of Texas Health Science Center, Houston; Claudia Pedroza, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (11):
- United States (11):
  - Indiana University College of Medicine, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Henry Ford Health System, Louisville, Kentucky
  - Rochester Regional Health, Rochester, New York
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Geisinger Health, Danville, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - Memorial Hermann Hospital System - Memorial City Medical Center, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Texas Health Science Center Houston with Memorial Hermann Hospital System - The Medical Center, Houston, Texas
  - Memorial Hermann Hospital System - The Woodlands Medical Center, The Woodlands, Texas

REFERENCES:
- [Derived] Chen PR, Artime CA, Sheth SA, Pedroza C, Ortega-Gutierrez S, Wolfe S, Sitton C, Kan P, Tanweer O, Chebl A, Schirmer CM, Morrow JT, Alderazi YJ, Bohnstedt B, Erkmen K, Samaniego EA, Garrido E, Savitz SI, Engstrom A, Aguilar E, Nguyen T, Barreto AD; SEGA Investigators. Sedation vs General Anesthesia for Endovascular Therapy in Acute Ischemic Stroke: The SEGA Randomized Clinical Trial. JAMA Neurol. 2025 Dec 1;82(12):1265-1273. doi: 10.1001/jamaneurol.2025.3775. PMID 41082222
- [Derived] Tosello R, Riera R, Tosello G, Clezar CN, Amorim JE, Vasconcelos V, Joao BB, Flumignan RL. Type of anaesthesia for acute ischaemic stroke endovascular treatment. Cochrane Database Syst Rev. 2022 Jul 20;7(7):CD013690. doi: 10.1002/14651858.CD013690.pub2. PMID 35857365

RESULTS

PARTICIPANT FLOW:
Groups:
- Sedation: The protocol does not specify a particular combination of drugs that must be used for sedation. The choice of specific drugs and dosages for achieving sedation will be up to the anesthesiologist.
  Sedation: The protocol does not specify a particular combination of drugs that must be used for sedation.
  The most common drugs utilized for sedation and wide dosing ranges are included in the protocol (i.e., sedation will be provided under the supervision of an anesthesiologist and may use a combination of fentanyl, midazolam, dexmedetomidine infusion (with or without loading dose), and/or low-dose propofol by intermittent bolus or infusion); however, the choice of specific drugs and dosages for achieving conscious sedation or general anesthesia will not be specified by the protocol but will be up to the anesthesiologist.
  Intra-arterial Thrombectomy: The first line therapeutic embolectomy device should be a stent retriever. Additional Endovascular therapies including, but not limited to, intra- or extracranial angioplasty ± stenting; antithrombotics (oral, IV or IA antiplatelets or anticoagulants) intra-arterial thrombolytics; are left to the decision of the local treatment team.
- General Anesthesia: General Anesthesia (GA): The protocol doesn't specify a particular combination of drugs that must be used for GA, the choice of drugs and dosages for achieving general anesthesia will not be specified by the protocol but will be up to the anesthesiologist.
  The most common drugs utilized for GA and wide dosing ranges included in the protocol are (GA will be provided under the supervision of an anesthesiologist and induction of anesthesia may be achieved with propofol and/or etomidate; muscle paralysis may be achieved with succinylcholine or non-depolarizing paralytic (rocuronium or vecuronium); and adjuvant lidocaine and fentanyl; if intravenous maintenance of anesthesia is used, it may be achieved by propofol infusion at 50 to 150 mcg/kg/min with redosing of non-depolarizing paralytic and fentanyl as needed; if inhalational maintenance of anesthesia is used it will be achieved with sevoflurane 1% to 2% or desflurane 3% to 6% end-tidal concentration with redosing of non-depolarizing paralytic and fentanyl as needed)
  Intra-arterial Thrombectomy: The first line therapeutic embolectomy device should be a stent retriever. Additional Endovascular therapies including, but not limited to, intra- or extracranial angioplasty ± stenting; antithrombotics (oral, IV or IA antiplatelets or anticoagulants) intra-arterial thrombolytics; are left to the decision of the local treatment team.
Period: Overall Study
Arm/Group | Sedation | General Anesthesia
Started | 130 | 130
Pass screening | 129 | 128
Completed | 120 | 120
Not Completed | 10 | 10

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were only collected for participants who were randomized and pass screening.
Groups:
- Total: Total of all reporting groups
Arm/Group | General Anesthesia | Sedation | Total
Number analyzed (Participants) | 128 | 129 | 257
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.9 (12.7) | 67.6 (13.8) | 66.77 (13.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 55 | 124
  Male | 59 | 74 | 133
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 21 | 44
  Not Hispanic or Latino | 98 | 100 | 198
  Unknown or Not Reported | 7 | 8 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 64 | 65 | 129
  Race: Black | 38 | 37 | 75
  Race: Asian | 3 | 2 | 5
  Race: More than one race | 7 | 7 | 14
  Race: Unknown | 16 | 18 | 34
Region of Enrollment [Number; unit: participants]
  United States | 128 | 129 | 257
Number of Participants who received intravenous tissue-type plasminogen activator treatment [Count of Participants; unit: Participants] | 78 | 72 | 150
Number of Participants with Atrial Flutter/Atrial Fibrillation [Count of Participants; unit: Participants] | 23 | 32 | 55
Number of Participants with a history of diabetes [Count of Participants; unit: Participants] | 26 | 34 | 60
Number of Participants with a History of Hypertension [Count of Participants; unit: Participants] | 77 | 95 | 172
Number of Participants with a History of Stroke [Count of Participants; unit: Participants] | 19 | 24 | 43
Number of Participants with Coronary artery disease [Count of Participants; unit: Participants] | 9 | 17 | 26
Number of Participants with Peripheral Vascular Disease [Count of Participants; unit: Participants] | 1 | 4 | 5
Number of participants with prior use of antiplatelets [Count of Participants; unit: Participants] | 26 | 36 | 62
Number of participants with prior use of anticoagulants [Count of Participants; unit: Participants] | 15 | 30 | 45
Vessels Occluded [Count of Participants; unit: Participants] — Participants can have more than one vessels occluded.
  Participants
    middle cerebral artery (MCA)- M1 | 77 | 69 | 146
    middle cerebral artery (MCA)- M2 Proximal | 30 | 33 | 63
    anterior cerebral artery (ACA)- A1 | 1 | 2 | 3
    anterior cerebral artery (ACA)- A2 Proximal | 1 | 1 | 2
    No Vessels Occluded | 6 | 9 | 15
    Unknown | 2 | 4 | 6
    Internal Carotid Artery (ICA) Terminus | 26 | 22 | 48
Time from Stroke Onset to Endovascular Therapy [Count of Participants; unit: Participants]
  less than 6 hours | 88 | 89 | 177
  6 hours to 16 hours | 40 | 40 | 80
Pre-stroke mRS [Count of Participants; unit: Participants] — The modified Rankin Scale (mRS) measures degree of disability/dependance after a stroke
  * 0: no symptoms/normal (physical, cognitive etc.)
  * 1: no significant disability despite symptoms; able to carry out all usual duties and activities
  * 2: slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance
  Participants
    0 | 102 | 105 | 207
    1 | 14 | 12 | 26
    2 | 12 | 12 | 24
Time from Stroke onset to Groin puncture [Median (Inter-Quartile Range); unit: minutes] — Population: Data were not collected from 56 participants in the general anesthesia arm and 65 participants in the sedation arm because the stroke onset was not witnessed, therefore the stroke onset time could not be collected.
  minutes
    number analyzed (Participants) | 72 | 64 | 136
    (all) | 488 [436 to 591] | 508 [445 to 602] | 495 [436 to 595]
Time from Door to Groin puncture [Median (Inter-Quartile Range); unit: minutes] — Population: Data were not collected from 6 participants in the general anesthesia arm because 3 were in-hospital patients, so door time can not be collected, and 3 participants did not receive Endovascular thrombectomy (EVT) procedure, so groin puncture time can not be collected. Data were not collected from 7 participants in the sedation arm because 3 were in-hospital patients, so door time can not be collected, and 4 did not undergo EVT procedure so, groin puncture time can not be collected.
  minutes
    number analyzed (Participants) | 122 | 122 | 244
    (all) | 78 [50 to 93] | 69 [52 to 93] | 71 [51 to 93]
Time from Angiosuite to Groin puncture [Median (Inter-Quartile Range); unit: minutes] — Population: Data were not collected from 3 participants in the general anesthesia arm because 3 participants did not receive Endovascular thrombectomy (EVT) procedure, so groin puncture time can not be collected. Data were not collected from 4 participants in the sedation arm because 4 participants did not undergo EVT procedure so, groin puncture time could not be collected.
  minutes
    number analyzed (Participants) | 125 | 125 | 250
    (all) | 17 [13 to 22] | 12 [9 to 19] | 15 [11 to 20]
Score on the National Institutes of Health Stroke Scale, or NIH Stroke Scale (NIHSS) [Median (Inter-Quartile Range); unit: score on a scale] — The National Institutes of Health Stroke Scale (NIHSS) is a tool used objectively quantify the impairment caused by a stroke. Total score ranges from 0 - 42, with a higher score indicating greater severity of impairment caused by stroke.
  0 No stroke symptoms 1-4 Minor stroke 5-15 Moderate stroke 16-20 Moderate to severe stroke 21-42 Severe stroke
  score on a scale | 15 [10 to 18] | 16 [11 to 20] | 15 [11 to 19]
Alberta Stroke Program Early CT Score [Median (Inter-Quartile Range); unit: score on a scale] — The Alberta Stroke Program Early CT Score (ASPECTS) is a 10-point quantitative topographic CT scan score used to assess the extent of ischemic changes in patients with acute middle cerebral artery (MCA) stroke. The score ranges from 0 to 10, with a higher score indicating less extensive early ischemic changes and a better prognosis. Population: Data were not collected from 3 participants in the general anesthesia arm and 1 participant in the sedation arm because CT imaging was not performed, therefore an ASPECT score could not be captured,
  score on a scale
    number analyzed (Participants) | 125 | 128 | 253
    (all) | 8 [7 to 10] | 9 [7 to 10] | 9 [7 to 10]

OUTCOME MEASURES:

1. Primary Outcome: Modified Ordinal Rankin Scale (mRS)
Description: mRS ranges from 0 to 6, with higher scores indicating greater disability. 6 categories are reported: number of participants who had a score of 0, 1, 2, 3, or 4 will be reported separately as 5 categories, and those who had a score of 5 or 6 will be combined and reported as a single category.
  0: no symptoms/normal (physical, cognitive etc.)
  1. no significant disability despite symptoms; able to carry out all usual duties and activities
  2. slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance
  3. moderate disability; requiring some help, but able to walk without assistance from another individual (use of walking aids alone is not counted as assistance)
  4. moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance
  5. severe disability; bedridden, incontinent and requiring constant nursing care and attention
  6. dead
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | General Anesthesia | Sedation
Number analyzed (Participants) | 120 | 120
Participants
  score of 0 | 16 | 11
  score of 1 | 21 | 23
  score of 2 | 20 | 13
  score of 3 | 21 | 24
  score of 4 | 9 | 16
  score of 5 or 6 | 33 | 33

2. Secondary Outcome: Dichotomized Modified Ordinal Rankin Scale (mRS)
Description: The modified Rankin Scale (mRS) ranges from 0 to 6, with higher scores indicating greater disability and where 0-2 is generally considered a good outcome with individuals assuming complete functional independence. 2 categories are reported: number of participants who had a score of 0-2, and number who had a score of 3-6.
  0: no symptoms/normal (physical, cognitive etc.)
  1. no significant disability despite symptoms; able to carry out all usual duties and activities
  2. slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance
  3. moderate disability; requiring some help, but able to walk without assistance from another individual (use of walking aids alone is not counted as assistance)
  4. moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance
  5. severe disability; bedridden, incontinent and requiring constant nursing care and attention
  6. dead
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | General Anesthesia | Sedation
Number analyzed (Participants) | 120 | 120
Participants
  Score of 0, 1, or 2 | 57 | 47
  Score of 3, 4, 5, or 6 | 63 | 73

3. Secondary Outcome: Number of Participants With Angiographic Reperfusion Defined as Modified a TICI Score of ≥ 2b
Description: The thrombolysis in cerebral infarction (TICI) grading system is a tool for determining the response of thrombolytic therapy for ischemic stroke. The TICI grade ranges from 0 to 3, with a higher score indicating greater perfusion.
  grade 0: no perfusion grade 1: penetration with minimal perfusion grade 2: partial perfusion grade 2A: only partial filling (less than two-thirds) of the entire vascular territory is visualized grade 2B: complete filling of all of the expected vascular territory is visualized but the filling is slower than normal grade 3: complete perfusion
Time Frame: post procedure within 6 hours
Population: Data were not collected from 6 participants in the general anesthesia arm and 7 participants in the sedation arm because they did not undergo the angiogram procedure.
Measure: Count of Participants; unit: Participants
Arm/Group | General Anesthesia | Sedation
Number analyzed (Participants) | 122 | 122
Participants | 118 | 116

4. Secondary Outcome: Score on the National Institutes of Health Stroke Scale, or NIH Stroke Scale (NIHSS)
Description: The National Institutes of Health Stroke Scale (NIHSS) is a tool used objectively quantify the impairment caused by a stroke. Total score ranges from 0 - 42, with a higher score indicating greater severity of impairment caused by stroke.
  0 No stroke symptoms 1-4 Minor stroke 5-15 Moderate stroke 16-20 Moderate to severe stroke 21-42 Severe stroke
Time Frame: 24-36 hours post procedure
Population: Data were not collected for 8 participants in the General Anesthesia arm and 5 participants in the Sedation arm because the National Institutes of Health Stroke Scale (NIHSS) assessment was not performed for these participants.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | General Anesthesia | Sedation
Number analyzed (Participants) | 120 | 124
score on a scale | 7 [3 to 14] | 6 [3 to 14]

5. Secondary Outcome: Number of Participants With Functional Independence as Indicated by an mRS Score of 0, 1, or 2
Description: The modified Rankin Scale (mRS) ranges from 0 to 6, with higher scores indicating greater disability and where 0-2 is generally considered a good outcome with individuals assuming complete functional independence.
  0: no symptoms/normal (physical, cognitive etc.)
  1. no significant disability despite symptoms; able to carry out all usual duties and activities
  2. slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance
  3. moderate disability; requiring some help, but able to walk without assistance from another individual (use of walking aids alone is not counted as assistance)
  4. moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance
  5. severe disability; bedridden, incontinent and requiring constant nursing care and attention
  6. dead
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | General Anesthesia | Sedation
Number analyzed (Participants) | 120 | 120
Participants | 57 | 47

6. Secondary Outcome: Quality of Life as Assessed by the European Quality of Life (EuroQol) 5 Dimensions 5 Level Version (EQ-5D-5L) Assessment
Description: The EQ-5D-5L score ranges from -0.59 to 1, where 1 is the best possible health state. Negative values represent health states perceived as worse than dead, which is equal to 0.
Time Frame: 90 days
Population: Data were not collected from 16 participants in the general anesthesia arm and Data were not collected from 14 participants in the Sedation arm because the European Quality of Life (EuroQol) 5 Dimensions 5 Level Version (EQ-5D-5L) assessment was not administered to these participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | General Anesthesia | Sedation
Number analyzed (Participants) | 112 | 115
score on a scale | 0.47 (0.44) | 0.46 (0.40)

7. Secondary Outcome: Number of Participants With Symptomatic Intracerebral Hemorrhage
Description: Symptomatic intracerebral hemorrhage was defined using the Safe Implementation of Thrombolysis in Stroke-Monitoring Study (SITS-MOST) definition, a ≥ 4 point increase in NIHSS score with a parenchymal hemorrhage type 2 within 36 hours.
Time Frame: 18-36 hours post procedure
Population: Data were not collected from 3 participants in the general anesthesia arm and Data were not collected from 4 participants in the Sedation arm because these participants did not undergo imaging at this timeframe therefore the data were not available for them.
Measure: Count of Participants; unit: Participants
Arm/Group | General Anesthesia | Sedation
Number analyzed (Participants) | 125 | 125
Participants | 1 | 3

8. Secondary Outcome: Number of Participants With All-cause Mortality
Time Frame: 18-36 hours post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | General Anesthesia | Sedation
Number analyzed (Participants) | 128 | 129
Participants | 11 | 9

9. Secondary Outcome: Number of Participants With Procedural Complications
Time Frame: 18-36 hours post procedure
Population: Data were not collected from 2 participants in the General Anesthesia arm and Data were not collected from 4 participants in the Sedation arm because the angiogram procedure was not performed.
Measure: Count of Participants; unit: Participants
Arm/Group | General Anesthesia | Sedation
Number analyzed (Participants) | 126 | 125
Participants | 4 | 5

10. Other Pre Specified Outcome: Time From Groin Puncture to Reperfusion
Time Frame: post procedure within 6 hours
Population: Data were not collected from 4 participants in the general anesthesia arm and 4 participants in the sedation arm because they did not undergo the EVT procedure.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | General Anesthesia | Sedation
Number analyzed (Participants) | 124 | 125
minutes | 41 [25 to 66] | 43 [29 to 65]

11. Other Pre Specified Outcome: Time From Door to TICI ≥ 2b Reperfusion
Time Frame: post procedure within 6 hours
Population: Data were not collected from 6 participants in the General Anesthesia arm and 6 participants in the Sedation arm because they did not have the EVT procedure.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | General Anesthesia | Sedation
Number analyzed (Participants) | 122 | 123
minutes | 121 [90 to 149] | 116 [93 to 138]

ADVERSE EVENTS:
Time Frame: from baseline to 90 days after discharge
Arm/Group | General Anesthesia | Sedation
All-Cause Mortality (participants affected / at risk) | 11/130 | 9/130
Serious Adverse Events (participants affected / at risk) | 62/130 | 65/130
Other Adverse Events (participants affected / at risk) | 0/130 | 0/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | General Anesthesia (N=130) | Sedation (N=130)
intracerebral hemorrhage asymptomatic (Vascular disorders) | 59 | 59
intracerebral hemorrhage symptomatic (Vascular disorders) | 1 | 3
Procedure Complications (Surgical and medical procedures) | 4 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-10): https://cdn.clinicaltrials.gov/large-docs/17/NCT03263117/Prot_SAP_001.pdf